CLINICAL TRIAL: NCT04577131
Title: Improving Adherence to Home Blood Pressure Monitoring With Pharmacist Support
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The tracker application has been withdrawn by developer and no other suitable tracker application has been identified to replace it.
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20019041
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- With check-ins (Experimental): Daily blood pressure monitoring with weekly check-ins
  Interventions: Behavioral: Weekly check-in
- Without check-ins (No Intervention): Daily blood pressure monitoring without weekly check-ins

INTERVENTIONS:
Behavioral: Weekly check-in — Weekly check-in phone calls from a pharmacist to review blood pressures and the number of times tested in that week
  Arms: With check-ins

SUMMARY:
The purpose of this research study is to evaluate the impact of monitoring blood pressure from home everyday with pharmacist support.

DETAILED DESCRIPTION:
High blood pressure is very common and increases risk of heart, kidney, brain, and eye disease. It is important to diagnose and treat high blood pressure to reduce risk of these complications. Getting blood pressure checked only when someone sees a doctor is not the best way to diagnose high blood pressure or to make sure blood pressure is well managed. Checking blood pressure at home gives a better idea of whether someone's blood pressure is normal or too high.

As part of their usual blood pressure monitoring, participants will be given an Omron 3 series or 5 series blood pressure monitor which has been cleared by the US Food and Drug Administration and validated to meet accuracy and performance requirements. For one month, participants will monitor their blood pressure once a day and then return the device to the clinic at the end of the study. Participants will text their blood pressure result to the American Heart Association's Check, Change, Control (CCC) secure online tracker.

As part of the research study, participants will also be randomized to either receive or not receive weekly check-in phone calls from a pharmacist to review their blood pressures and the number of times they tested in that week. Approximately 50 individuals will participate in this study. Participation in this study will last 1 month.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Uncontrolled hypertension (BP > 130/80 mm Hg)

Exclusion Criteria:

* non-English speaking patients
* patients without a mobile phone or texting capability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Change in adherence to home blood pressure monitoring | 1 month
  Proportion of days blood pressure is measured based on data from the blood pressuring monitor
Change in proportion of participants with a blood pressure <130/80 mm Hg. | 1 month
  Proportion of participants with a blood pressure <130/80 mm Hg.

CONTACTS AND LOCATIONS:
Overall Officials: Dave Dixon, PharmD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No